CLINICAL TRIAL: NCT02906696
Title: An Open-Label Phase II Dose Optimization Study of Bosutinib at a Starting Dose of 300 Mg Daily for Adult Patients With Chronic Myeloid Leukemia (CML) in Chronic Phase Post Frontline TKI Failure
Brief Title: Bosutinib in Treating Patients With Chronic Myeloid Leukemia in Chronic Phase After Frontline TKI Failure
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated per PI's request due to competing priorities.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-0081; NCI-2016-01954 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2016-0081 (Other: M D Anderson Cancer Center); P30CA016672 (NIH)
Record Dates: First submitted 2016-09-15; First posted 2016-09-20 (Estimated); Results first posted 2020-04-22 (Actual); Last update posted 2020-05-11 (Actual); Status verified 2020-04

CONDITIONS: Blasts Under 15 Percent of Bone Marrow Nucleated Cells; Blasts Under 15 Percent of Peripheral Blood White Cells; Blasts Under 30 Percent of Bone Marrow Nucleated Cells; Blasts Under 30 Percent of Peripheral Blood White Cells; Chronic Phase Chronic Myelogenous Leukemia, BCR-ABL1 Positive
MeSH Terms: conditions — Leukemia, Myeloid, Chronic-Phase | interventions — bosutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (bosutinib) (Experimental): Patients receive bosutinib PO daily on days 1-28. Cycles repeat every 28 days for up to 2 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Bosutinib; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Bosutinib — Given PO
  Other Names: Bosulif; SKI 606; SKI-606
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase II trial studies how well bosutinib works in treating patients with chronic myeloid leukemia in chronic phase after frontline tyrosine kinase inhibitor (TKI) failure. Bosutinib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the response rate within 24 weeks in patients in chronic phase receiving bosutinib with the starting dose of 300 mg per day, with potential escalation to 400 mg, 500 mg and 600 mg per day.

SECONDARY OBJECTIVES:

I. Safety of dosing schedule. II. Frequency of treatment interruptions and dose reductions. III. Determine the rate of BCR-ABL/ABL < 10% at 3 months and < 1% at 6 months on the international scale and the rate of complete cytogenetic response (CCyR) at 6 months after the start of treatment.

IV. Determine the cumulative rate of CCyR. V. Determine the rate of major molecular response, molecular response (MR)4, MR4.5 and complete molecular response.

VI. Determine long-term outcomes, including progression-free survival, event-free survival, and overall survival.

VIII. Investigate the correlation between ABL kinase domain mutations, if present at the time of enrollment, with outcome.

IX. Determine the rate of development and type of ABL kinase domain mutations during therapy with bosutinib.

OUTLINE:

Patients receive bosutinib orally (PO) daily on days 1-28. Cycles repeat every 28 days for up to 2 years in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 12 weeks for up to 2 years, every 24 weeks for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic myeloid leukemia (CML) in chronic phase who have resistance and/or intolerance to frontline TKI therapy; resistance is defined as lack (lack defined as response not achieved or lost by the given dates mentioned hereafter) of CHR (complete hematologic response) within 3 months, lack of major cytogenetic response (MCyR) within 6 months, and lack of CCyR within 12 months of therapy with frontline TKIs; in addition, loss of MCyR, CCyR or MMR at any time during the course of therapy is also considered resistance to therapy; intolerance is defined as persistent or severe toxicity that is unacceptable to the patient
* Chronic phase disease is defined as:

  * < 15% blasts in peripheral blood and bone marrow;
  * < 30% blasts plus promyelocytes in peripheral blood and bone marrow;
  * < 20% basophils in peripheral blood;
  * >= 100 x 10^9/L platelets (>= 100,000/mm^3);
  * No evidence of extramedullary disease except hepatosplenomegaly; and
  * No prior diagnosis of accelerated phase (AP) or blastic phase-chronic myeloid leukemia (BP-CML); patients with clonal evolution but no other criteria for accelerated phase are eligible
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
* Creatinine less than or equal to 2.0 mg/dl
* Bilirubin less than or equal to 2.0 mg/dl
* Alanine aminotransferase (ALT) less than or equal to 3 times institutional upper limit of normal
* Females of childbearing potential must have a negative serum or urine beta human chorionic gonadotrophin (beta-hCG) pregnancy test result within 14 days prior to the first dose of study drugs and must agree to use one of the following effective contraception methods during the study and for 30 days following the last dose of study drug; effective methods of birth control include:

  * Birth control pills, shots or implants (placed under the skin by a health care provider) or patches (placed on the skin);
  * Intrauterine devices (IUDs);
  * Condom or occlusive cap (diaphragm or cervical/vault caps) used with spermicide; females of non-childbearing potential are those who are postmenopausal greater than 1 year or who have had a bilateral tubal ligation or hysterectomy
* Males who have partners of childbearing potential must agree to use an effective contraceptive method during the study and for 30 days following the last dose of study drug
* Patients or their legally authorized representative must provide written informed consent

Exclusion Criteria:

* Women who are pregnant or lactating
* Known to be human immunodeficiency virus (HIV)+
* Active and uncontrolled disease/infection that in the opinion of the treating physician and principal investigator may affect the ability to participate in the trial or put the patient at unduly high risk
* Unable or unwilling to sign the informed consent document
* Received no other investigational therapy within the past 14 days
* Presence of T315I mutation by ABL1 sequencing
* Patient is currently in complete cytogenetic remission (CCyR)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2016-10-28 (Actual); Primary Completion 2019-08-08 (Actual); Study Completion 2019-08-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip A Thompson, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: October 2016 to November 2018
Period: Overall Study
Arm/Group | Treatment (Bosutinib)
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Bosutinib)
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 2
Age, Continuous [Median (Full Range); unit: years] | 44 [41 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Response Rate
Description: Response is defined as follows: 1) For patients who do not currently have a partial cytogenetic response (PCyR), achievement of major cytogenetic response is considered a response. 2) For patients who are currently in PCyR, achievement of CCyR is considered a response. The Simon's optimal two-stage design will be used for interim futility monitoring. Will be estimated along with the 95% credible interval.
Time Frame: Up to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Bosutinib)
Number analyzed (Participants) | 8
Participants | 6

2. Secondary Outcome: Number of Participants With Treatment Interruptions and Dose Reductions
Description: Will be summarized.
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Bosutinib)
Number analyzed (Participants) | 8
Participants
  Interruptions | 6
  Reductions | 4

3. Secondary Outcome: Rates of Major Molecular Response (MR), MR4, MR4.5 and Complete Molecular Response
Description: Will be estimated along with the exact 95% confidence intervals. Molecular assessments are based on quantitative reverse transcriptase polymerase chain reaction for Bcr-Abl in peripheral blood. Molecular response is categorized as MMR (Bcr-Abl/Abl ratio of </= 0.1% in the international scale), MR4 (Bcr-Abl/Abl </= 0.01%), and MR4.5 (BCR-ABL/ABL </=0.0032%).
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Bosutinib)
Number analyzed (Participants) | 8
Participants
  Complete Molecular Response (CMR) | 2
  MR4.5 | 3
  MR4 | 3
  Major Molecular Response (MMR) | 5

4. Secondary Outcome: Rates of BCR-ABL/ABL <10%
Description: Will be assessed using the international scale. Will be estimated along with the exact 95% confidence intervals.
Time Frame: At 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Bosutinib)
Number analyzed (Participants) | 8
Participants | 3

5. Secondary Outcome: Rates of BCR-ABL/ABL < 1%
Description: Will be assessed using the international scale. Will be estimated along with the exact 95% confidence intervals.
Time Frame: At 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Bosutinib)
Number analyzed (Participants) | 8
Participants | 2

6. Secondary Outcome: Overall Survival
Description: Will be assessed by Kaplan-Meier methods. Cox proportional hazards regression models will be fit to assess the association between patient characteristics including survival outcome. Time from date of treatment start until date of death due to any cause or last Follow-up.
Time Frame: Up to 2 years
Measure: Median (Full Range); unit: Months
Arm/Group | Treatment (Bosutinib)
Number analyzed (Participants) | 8
Months | 20.26 [13.63 to 22.90]

7. Secondary Outcome: Event-free Survival
Description: Time from date of treatment start until the date of first objective documentation of disease-relapse.
Time Frame: Up to 2 years
Measure: Median (Full Range); unit: Months
Arm/Group | Treatment (Bosutinib)
Number analyzed (Participants) | 8
Months | 13.97 [3.06 to 22.90]

8. Secondary Outcome: Transformation-free Survival
Description: Will be assessed by Kaplan-Meier methods. Transformation-free survival is defined as the time from treatment initiation until either progression to AP/BP or death from any cause.
Time Frame: Up to 2 years
Measure: Median (Full Range); unit: Months
Arm/Group | Treatment (Bosutinib)
Number analyzed (Participants) | 8
Months | 13.97 [3.75 to 22.90]

9. Secondary Outcome: Change of ABL Kinase Domain Mutation Status
Description: Will be summarized and its association with survival outcomes will be analyzed through landmark analyses. Cox proportional hazards regression models will be fit to assess the association between patient characteristics including ABL kinase domain mutation status.
Time Frame: Baseline up to 2 years
Population: There were not any at the start of treatment so there were not any mutation status to follow. These were not done.
Arm/Group | Treatment (Bosutinib)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: up to 2 years
Arm/Group | Treatment (Bosutinib)
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 4/8
Other Adverse Events (participants affected / at risk) | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Bosutinib) (N=8)
Chest Pain (Cardiac disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Gastrointestinal Bleed (Gastrointestinal disorders) | 1 (1)
Arterial Rupture (Injury, poisoning and procedural complications) | 1 (1)
Viral Infection (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Bosutinib) (N=8)
Abdominal Pain (General disorders) | 2 (2)
Elevated Alanine transaminase (Investigations) | 4 (11)
Angioedema (Blood and lymphatic system disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Aspartate transaminase (Investigations) | 2 (4)
Bruising (Injury, poisoning and procedural complications) | 1 (1)
Chest Pain (General disorders) | 1 (1)
Elevated Creatinine (Investigations) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 7 (7)
Fatigue (General disorders) | 5 (5)
Fever of Unknown origin (General disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Headache (General disorders) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Irregular Menstration (Reproductive system and breast disorders) | 1 (1)
Mucositis (Gastrointestinal disorders) | 1 (1)
Sodium (Metabolism and nutrition disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Sensory Neuropathy (Nervous system disorders) | 1 (1)
Periorbital Edema (Eye disorders) | 1 (1)
Pruritis (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 3 (3)
Upper Respiratory Infection (Infections and infestations) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Yeast Infection (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-20): https://cdn.clinicaltrials.gov/large-docs/96/NCT02906696/Prot_SAP_000.pdf